CLINICAL TRIAL: NCT03894982
Title: Family Learning on Asthma Topics
Acronym: FLOAT
Status: Completed | Type: Observational
Sponsor: University of Colorado, Denver (Other)
Responsible Party: Sponsor
Other Study IDs: 19-0442
Record Dates: First submitted 2019-03-27; First posted 2019-03-29 (Actual); Last update posted 2020-08-04 (Actual); Status verified 2020-07

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Observational Model: Family Based | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- What is Asthma: Reviewing asthma is a lung disease. There is no cure, but asthma can be well controlled so that your child can be healthy and join in all their favorite activities.
  Asthma causes the airways (breathing tubes in the lungs) to get smaller, making it hard to breathe.Common symptoms of asthma are coughing, wheezing, chest tightness and trouble breathing.
  These symptoms are ongoing and get better with asthma medicines.
  Interventions: Other: Group Classes
- Triggers: Reviewing specifics around children with asthma have extra sensitive airways and many things around them can make their asthma worse. The things around your child that cause an asthma attack are called triggers. Triggers are different for each child. Your doctor can help you figure out your child's triggers. Try to keep your child away from their triggers, especially at home and at school where your child spends most of their time.
  Interventions: Other: Group Classes
- Medications and Asthma Action Plan: Review what is an asthma action plan, how to use an asthma action and the medications listed on each individuals plan.
  Interventions: Other: Group Classes

INTERVENTIONS:
Other: Group Classes — Family Learning on Asthma Topics classes will aim to emphasize, encourage, and support teaching methods that include standardized instructions. There will be three topics lasting approximately 45 minutes: General Asthma Knowledge; Asthma Triggers, Medications, and Self-Management. These topics were chosen based on the EPR-3 guideline recommendations to ensure the continuity of messaging. Each class size will be approximately 8 persons and will be taught by a Certified Asthma Educator (AE-C) and will be held in the Family Learning Center at the Children's Hospital Colorado. Classes will be taught in both English and Spanish.

SUMMARY:
1. Hypothesis: The Family Learning on Asthma Topics (F.L.O.A.T) in the form of a a group teaching environment for family education stemming from standardized education materials on asthma, created and taught by nationally certified asthma educators will promote optimal asthma knowledge, management and quality of life among the individuals with asthma and their caregivers.
2. Aim 1: To determine if the availability of educational services outside of regular clinic hours or admission status could improve asthma outcomes and decrease unnecessary medical utilization.
3. Aim 2: By providing small-group learning environments for families, the investigators aim to encourage families to learn from each other's experiences and to decrease stigma around the disease.

DETAILED DESCRIPTION:
I. Hypotheses and Specific Aims:

1. Hypothesis: The Family Learning on Asthma Topics (F.L.O.A.T) in the form of a a group teaching environment for family education stemming from standardized education materials on asthma, created and taught by nationally certified asthma educators will promote optimal asthma knowledge, management and quality of life among the individuals with asthma and their caregivers.
2. Aim 1: To determine if the availability of educational services outside of regular clinic hours or admission status could improve asthma outcomes and decrease unnecessary medical utilization.
3. Aim 2: By providing small-group learning environments for families, the investigators aim to encourage families to learn from each other's experiences and to decrease stigma around the disease.

II. Background and Significance:

Despite recent improvements in treatment and the ongoing research in better understanding of the disease, emergency room visits and hospitalization rates for asthma remain high. The Centers for Disease Control and Prevention surveillance data reports that at a national level, health care use for emergency department services for asthma was 1.6 million in 2013, and that of 439,435 hospital admissions for asthma 136,669 or 31% are for children below the age of 18 years of age. The annual cost of asthma on the U.S. economy equates to more than $80 billion in medical expenses, including days missed from school, work and even death. Nurmagambetov, et.al. in their study state that the "combined costs of medical care, mortality, and absenteeism render the total cost of asthma a substantial and serious economic burden on society. These findings highlight the critical need to support and further strengthen asthma control strategies through increased provision of guideline-based care, improvements in self-management, and reduction of environmental asthma triggers to reduce ER visits, hospitalizations, absenteeism, and mortality".

Bäuerle et al. used a prospective single-center controlled trial to show that by providing motivating and patient-oriented didactics on asthma, there is a statistically significant increase in asthma health outcomes and that asthma control can be improved by education measures. Although it is a key component of all international asthma guidelines, education in self-management is still insufficiently available in primary care settings. In the ambulatory setting, there are some families that require more extensive education and time is limited in a usual care appointment to address all their specific asthma needs.

Providing patient education by an experienced asthma educator is an important step in supporting patients and families as they are diagnosed with asthma and as they adapt to life with a chronic condition. Educating families about the nature of the disease, triggers, identification of early signs and symptoms, principles of treatment, and asthma management can reduce children's use of acute care services. According to Srof et al., asthma management education programs should be connected to the chronic illness management within the fabric of the family system. The paradigm of group education supports engagement, promoting communication among all participants including facilitator to enhance a social construct for validating personal experiences, empowering caregivers, and solving asthma management problems.

III. Preliminary Studies/Progress Report: none

IV. Research Methods

A. Outcome Measure(s):

Decrease emergency room visits, hospitalizations, and systemic steroid use for each child 12 months after completing the three, group classroom educational sessions.

1. Description of Population to be Enrolled:

   The investigators will enroll legal guardians and or primary caregiver (18 years and older) of children 4-17 years of age along with those children/adolescents who have a diagnosis of asthma, and have documented poor control as evidenced by requiring two or more systemic steroids, one or more hospitalizations and/or two or more ED visits due to asthma in the 12 months prior to the asthma clinic or hospital visit. Patients and caregivers will be English or Spanish speaking.
2. Study Design and Research Methods:

   Patients and caregivers will be recruited from the Pulmonary outpatient clinic and inpatient services at Children's Hospital Colorado. Patients will also be referred to the Family Learning on Asthma Topic (F.L.O.A.T) program by health care providers participating in these clinics/inpatient service. Children will be: 1) 4-17 years age, 2) have poor evidence of asthma control based on > 2 systemic steroid courses; > 2 Emergency Room visits; and >1 hospitalization for asthma exacerbation in the preceding 12 months. The investigators anticipate to enroll 75 patients and enrollment to begin in the Spring 2019 through the Spring 2020.

   Family Learning on Asthma Topics classes will aim to emphasize, encourage, and support teaching methods that include standardized instructions. There will be three topics lasting approximately 45 minutes: General Asthma Knowledge; Asthma Triggers, Medications, and Self-Management. These topics were chosen based on the EPR-3 guideline recommendations to ensure the continuity of messaging. Each class size will be approximately 8 persons and will be taught by a Certified Asthma Educator (AE-C) and will be held in the Family Learning Center at the Children's Hospital Colorado. Classes will be taught in both English and Spanish. An in person Spanish asthma educator will be available to help teach the classes.

   The materials used for each class were created by the CHCO Health Literacy Team in collaboration with Asthma Educator Certified members of the Breathing Institute to ensure that evidence-based information will be communicated effectively to patients and families. Instead of a lecture style course, each class will facilitate interactive learning for patients and families to help them prepare for real life problem-solving and to promote self-awareness regarding medication use.

   Patient and families enrolled will be notified of the class schedule and receive reminders 1 week and the day before each of their classes either through email, phone call and or text messaging.

   There will be a general asthma knowledge questionnaire consisting of 12 questions and the standardized Asthma Control Test (ACT) that consists of 7 standardized questions, one for children 4 - 11 years of age and one for children 12 years and older, that participants will fill out at the start of their first class. After each class, there will be 4 questions to be answered regarding their understanding of that class. Handouts and visuals will be available in English and Spanish pertaining to information about that class. Other class materials will include a folder to keep their handouts in and paper and pencils for note taking. Peak flow meters and their Asthma Action Plans will also be provided. At the completion of the class series there will be a satisfaction survey, participants will fill out anonymously.

   Twelve months following the completion of the class series, the investigators will be conducting a chart review gathering data on frequency of emergency room visits, hospitalizations and systemic steroid use for asthma exacerbations along with any routine follow up visits for asthma.
3. Description, Risks and Justification of Procedures and Data Collection Tools:

Data collected will be through pre and post class questionnaires, Asthma Control Test (ACT), validated Inhaler Technique Assessment Tool (iDAT), and demographic information filled out by the families and noted in their EMR (EPIC). Information about participant's asthma care utilization and systemic steroid use will be obtained through EMR/EPIC chart review, 12 months prior to enrollment and 12 months post last completed class. All information will be entered in to a secure REDCap data base and paper copies will be kept in the locked research cabinet of study personnel.

E. Potential Scientific Problems: The investigators do not anticipate any scientific problems

F. Data Analysis Plan:

Inclusion requirements will be defined through the electronic medical record based on inclusion requirements by either the outpatient pulmonary team or inpatient asthma education team.

After enrollment the following information will be placed into RedCap (HIPPA compliant database) from the EMR: Childs name, DOB, Race, Ethnicity, Cell phone number, Email, Zip Code, Sex, Preferred language (caregiver), Pulmonary or Allergy specialist seen within the previous year, Payer, Hospital visits (ED and hospital visits) 12 months prior to consent.

Right after enrollment a pre-knowledge base survey of 12 questions and asthma control survey of 7 questions will be sent via RedCap to caregivers defined phone and email. The data will be collected electronically and stored in RedCap.

Throughout the 4-month study period, every week an administrative support person will pull the child's name, caregivers name, designated contact phone number, and email from RedCap databased to send a text, email, and phone call reminders of upcoming classes and asking the caregiver to reply electronically if they are planning on attending. The administrative assistant will review the reply's and notify the educators of the number of class attendees and their names.

Upon completing each of the three classes the instructor will ask for the administrative assistant to send a post knowledge bases survey of 4 questions out of RedCap to the primary caregiver. The electronic responses will be electronically entered into RedCap.

Upon completion of the 3 classes and/or 4months the administrative assistant will send a post-knowledge survey consisting of 12 questions, an asthma control test survey of 7 questions, and a satisfaction survey to the primary caregiver. The electronic responses will be entered into RedCap.

Each quarter the overview of pre-knowledge base survey results, post-knowledge survey results and satisfaction survey will be reviewed by the team members to evaluate if any changes need to be made to the education curriculum.

Child specific data will be reviewed 12 months after completion of the classes and/or study.

G. Summarize Knowledge to be Gained:

By conducting this group focused asthma education series for high risk asthmatics and their care givers, the investigators anticipate improved knowledge along with retention of knowledge gained through these classes thereby reducing exacerbations, and need for acute care interventions. Group centered learning will enhance opportunities to learn from others who may have similar experiences and will generate discussion and new skills and ideas.

ELIGIBILITY:
Inclusion Criteria:

* Legal guardians and or primary caregiver (18 years and older) of children 4-17 years of age
* Children/adolescents who have a diagnosis of asthma, and have documented poor control as evidenced by requiring two or more systemic steroids, one or more hospitalizations and/or two or more ED visits due to asthma in the 12 months prior to the asthma clinic or hospital visit.
* Patients and caregivers will be English or Spanish speaking.

Exclusion Criteria:

* children < 4 yrs of age
* children with multiple chronic lung diseases
* Children and families whose primary language is other than English or Spanish

Ages: 4 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Despite recent improvements in treatment and the ongoing research in better understanding of the disease, emergency room visits and hospitalization rates for asthma remain high, with 31% of these visits are children below the age of 18 years of age.
  Providing patient education by an experienced asthma educator is an important step in supporting patients and families as they are diagnosed with asthma and as they adapt to life with a chronic condition. Educating families about the nature of the disease, triggers, identification of early signs and symptoms, principles of treatment, and asthma management can reduce children's use of acute care services.
Sampling Method: Probability Sample
Enrollment: 10 (Actual)
Dates: Start 2019-05-05 (Actual); Primary Completion 2020-05-31 (Actual); Study Completion 2020-05-31 (Actual)

PRIMARY OUTCOMES:
Change the number of hospital visits of participants with asthma | 12 months from completion of the classroom sessions
  Change the number of hospital visits of participants with asthma through comprehensive asthma education
Change the number of emergency room or urgent care visits of participants with asthma | 12 months from completion of the classroom sessions
  Change the number of emergency room or urgent care visits of participants with asthma through comprehensive asthma education
Change the amount of oral steroids taken by the participants for asthma exacerbations | 12 months from completion of the educational sessions
  Change the amount of oral steroids taken by participants for asthma exacerbation through comprehensive asthma education

CONTACTS AND LOCATIONS:
Overall Officials: Stan Szefler, MD, Principal Investigator — Children's Hospital Colorado
Locations (1):
- Children's Hospital Colorado, Aurora, Colorado, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] CDC - Asthma - Data and Surveillance - Asthma Surveillance Data. (2016, September 8). Retrieved from https://www.cdc.gov/asthma/asthmadata.htm
- [Background] Nurmagambetov T, Kuwahara R, Garbe P. The Economic Burden of Asthma in the United States, 2008-2013. Ann Am Thorac Soc. 2018 Mar;15(3):348-356. doi: 10.1513/AnnalsATS.201703-259OC. PMID 29323930
- [Background] Bauerle K, Feicke J, Scherer W, Sporhase U, Bitzer EM. Evaluation of a standardized patient education program for inpatient asthma rehabilitation: Impact on patient-reported health outcomes up to one year. Patient Educ Couns. 2017 May;100(5):957-965. doi: 10.1016/j.pec.2016.11.023. Epub 2016 Nov 28. PMID 27993435
- [Background] Boulet LP, Boulay ME, Gauthier G, Battisti L, Chabot V, Beauchesne MF, Villeneuve D, Cote P. Benefits of an asthma education program provided at primary care sites on asthma outcomes. Respir Med. 2015 Aug;109(8):991-1000. doi: 10.1016/j.rmed.2015.05.004. Epub 2015 May 14. PMID 26162708
- [Background] Srof B, Taboas P, Velsor-Friedrich B. Adolescent asthma education programs for teens: review and summary. J Pediatr Health Care. 2012 Nov-Dec;26(6):418-26. doi: 10.1016/j.pedhc.2011.03.010. Epub 2011 May 12. PMID 23099308
- [Background] McCarty K, Rogers J. Inpatient asthma education program. Pediatr Nurs. 2012 Sep-Oct;38(5):257-62, 269; quiz 263. PMID 23189776
- [Background] National Heart Lung and Blood Institute (US). Expert Panel Report 3: Guidelines for the Diagnosis and Management of Asthma Clinical Practice Guidelines National Asthma Education and Prevention Program, Third Expert Panel on the Diagnosis and Management of Asthma. http://www.nhlbi.nih. gov/guidelines/asthma/asthgdln.htm (Accessed March 19 2018).